CLINICAL TRIAL: NCT03567967
Title: The EValuating Interventions in Diabetogenic Environments Through Natural Controlled Experiments (EVIDENCE) Trial
Brief Title: Fruit and Vegetable Vouchers With and Without an SSB Tax
Acronym: EVIDENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 43831
Record Dates: First submitted 2018-05-31; First posted 2018-06-26 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Diseases
Keywords: nutrition; fruits and vegetables; sugar-sweetened beverages
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fruit

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: 24-hour dietary recalls are conducted by blinded registered dietitians
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- San Francisco (Experimental): Each study participant will receive four paper vouchers per month for a total of six months. Each of these vouchers can be redeemed for fresh or frozen fruits and vegetables at a number of specified local corner stores, supermarkets, or farmer's markets. The San Francisco participants will receive and spend these vouchers in an environment which has implemented a sugar-sweetened beverage tax.
  Interventions: Behavioral: Fruit and vegetable voucher
- Los Angeles (Active Comparator): Each study participant will receive four paper vouchers per month for a total of six months. Each of these vouchers can be redeemed for fresh or frozen fruits and vegetables at a number of specified local corner stores, supermarkets, or farmer's markets. The Los Angeles participants will receive and spend these vouchers in an environment which has NOT implemented a sugar-sweetened beverage tax.
  Interventions: Behavioral: Fruit and vegetable voucher

INTERVENTIONS:
Behavioral: Fruit and vegetable voucher — Participants will receive four vouchers, each dated for a month, to be used on fruits and vegetables at specified local corner stores, supermarkets, and farmer's markets for a duration of six months. Each study participant will have the same intervention, as this is a non-inferiority trial to compare voucher use in LA and test whether the nutritional effects of that use are non-inferior to use in SF.
  Other Names: Voucher

SUMMARY:
We aim to examine whether a purchasing incentive for healthy foods has the same effect on dietary intake in a community with and a community without a purchasing penalty for unhealthy foods. We will perform a randomized non-inferiority trial in two locations, San Francisco (SF) and Los Angeles (LA) to test whether a voucher for purchasing fresh fruits and vegetables has a similar effect in LA and in SF, where the former does not but the latter does have a tax on sugar-sweetened beverages. Participants will be recruited from 4 neighborhoods (N=312) with 2 SF neighborhoods (exposed to the SSB tax) and 2 LA neighborhoods (not exposed to the SSB tax).

DETAILED DESCRIPTION:
We will test the hypothesis that a positive incentive for healthy foods (fresh fruits and vegetables, F&Vs) will be utilized as effectively in a community without a purchasing penalty for unhealthy foods (a sugar-sweetened beverage [SSB] tax) as in a community with a purchasing penalty for unhealthy foods (a SSB tax). Our experiment will test the empirically-driven hypothesis in a real-world setting through a noninferiority design: comparing the impact of F&V vouchers in two counties, one without (Los Angeles) and one with (San Francisco) a SSB tax.

Each study participant will receive four paper vouchers per month for a total of six months. Each of these vouchers can be redeemed for fresh or frozen fruits and vegetables at a number of specified local corner stores, supermarkets, or farmer's markets.

Half of these participants will receive and spend these vouchers in an environment which has implemented a SSB tax (SF); the other half will receive and spend these same vouchers in a non-tax environment (LA).

Each individual participant will be enrolled in the study for a total of seven months from initial orientation and participant consent (M0) to final data collection during final month of intervention (M6).

We are using a non-inferiority trial design. We are aiming to test whether there is a significant difference in total cup-equivalents of F&V intake in LA participants as compared to SF participants when given F&V vouchers. That is, we aim to test whether the F&V voucher is less effective in LA than in SF. This is important to test because it has been purported that SF has a unique food environment with high accessibility to fresh F&V through farmer's markets and a plethora of corner stores, as well as a SSB tax that discourages less healthy foods, potentially leaving more funds for healthier F&Vs. Thus, we aim to determine the change in consumption of F&V in LA participants is non-inferiority to that of SF participants, when both are given F&V vouchers.

ELIGIBILITY:
Inclusion Criteria:

1. Understand English sufficiently to provide informed consent;
2. Provision of signed and dated informed consent form;
3. Stated willingness to comply with all study procedures and availability for the duration of the study;
4. Any gender, aged 21 years or older;
5. Have self-reported income ≤250% of the federal poverty level;
6. Have regular access to a mobile phone;
7. Have a safe and secure mailing address at which to receive vouchers;
8. Be a resident of the Counties of San Francisco or Los Angeles as defined by official municipal boundaries.

Exclusion Criteria:

1. Currently participating in any other dietary or nutrition study that would impact his or her normal eating patterns;
2. Currently be enrolled in and receiving EatSF, CHIVES, or Vouchers4Veggies vouchers;
3. Has active diagnosis of cancer or congestive heart failure;
4. Is planning to move out of San Francisco or Los Angeles in the next 12 months;
5. Currently pregnant.
6. Currently live with and share a food budget with a current Vouchers4Veggies, EVIDENCE, or CHIVES study participant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Change in fruit and vegetable consumption | Month 0 to Month 6
  Change in fruit and vegetable consumption from baseline (BL), i.e., before voucher receipt, to the end of the intervention at the end of month 6 (M6), i.e., during the final month of voucher receipt, measured by two 24-hour recalls at each data collection point (BL and M6).

SECONDARY OUTCOMES:
Change in nutrition quality per HEI score | Month 0 to Month 6
  Change in nutrition quality of study participants from BL to M6, measured by the Healthy Eating Index (HEI), which is calculated from two 24-hour recalls at each data collection point (BL and M6).
Change in nutrition quality per AHEI score | Month 0 to Month 6
  Change in nutrition quality of study participants from BL to M6, measured by the Alternative Healthy Eating Index (AHEI), which is calculated from two 24-hour recalls at each data collection point (BL and M6).
Change in SSB consumption | Month 0 to Month 6
  Change in SSB consumption from BL to M6, measured in change in fluid ounces, as measured by two 24-hour recalls at each data collection point (BL and M6).
Change in overall caloric intake | Month 0 to Month 6
  Change in overall caloric intake from BL to M6, measured in change in kcal, as measured by two 24-hour dietary recalls at each data collection point (BL and M6).
Overall percentage of vouchers redeemed | Month 0 to Month 6
  Overall percentage of vouchers redeemed per participant, measured by how many vouchers each participant redeemed as compared to how many vouchers they received over the 6 month intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Basu, MD, PhD, Principal Investigator — Assistant Professor of Medicine; Dean Schillinger, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: San Francisco program — https://is.gd/chivesprojectSF
- See also: Los Angeles program — https://is.gd/chivesprojectLA